CLINICAL TRIAL: NCT04686136
Title: A Phase 3, Multicenter, Open-Label 156-Week Extension Study To Evaluate The Long-Term Safety And Tolerability Of Oral Atogepant For The Prevention Of Migraine In Participants With Chronic Or Episodic Migraine
Brief Title: A Long-Term Safety and Tolerability Extension Study Evaluating Atogepant for the Prevention of Chronic or Episodic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3101-312-002; 2020-002470-27 (EudraCT Number)
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Episodic Migraine; Chronic Migraine
Keywords: Episodic migraine; Chronic migraine
MeSH Terms: interventions — atogepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atogepant 60 mg (Experimental): Taken once daily
  Interventions: Drug: Atogepant 60 mg

INTERVENTIONS:
Drug: Atogepant 60 mg — Tablets containing 60 mg of Atogepant

SUMMARY:
This study will evaluate the Long-Term Safety and Tolerability of Atogepant 60 mg daily for the Prevention of Migraine in Participants with Chronic or Episodic Migraine

ELIGIBILITY:
Inclusion Criteria:

- Eligible participants who completed Visit 7, and Visit 8 if applicable, of Study 3101-303-002 or Study 3101-304-002 without significant protocol deviations and who did not experience an Adverse Event that may indicate an unacceptable safety risk.

Exclusion Criteria:

* Participants requiring any medication, diet, or nonpharmacological treatment on the list of prohibited concomitant medications or treatments that cannot be discontinued or switched to an allowable alternative.
* Participants with an ECG indicating clinically significant abnormalities at Visit 1.
* Participants with hypertension at Visit 1.
* Participants with a significant risk of self-harm, or of harm to others; participants who report suicidal ideation with intent, with or without a plan, since the last visit, must be excluded.
* Participants with clinically significant hematologic, endocrine, cardiovascular, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with at Least 1 Treatment Emergent Adverse Event | 156 weeks

SECONDARY OUTCOMES:
Percentage of Participants with Clinically Significant Laboratory Values (Chemistry, Hematology, Urinalysis) as assessed by the Investigator | 156 weeks
Percentage of Participants with Clinically Significant Electrocardiograms (ECGs) Findings as assessed by the Investigator | 156 weeks
Percentage of Participants with Clinically Significant Vital Sign Measurements as assessed by the Investigator | 156 weeks
Columbia-Suicide Severity Rating Scale (C-SSRS) Assessing Suicidal Ideation and Behaviour using 5-Point Scales | 156 weeks
  A clinician-rated instrument that reports the severity of both suicidal ideation and behavior. Suicidal ideation is classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 5-item scale: 0 (no suicidal behavior), 1 (preparatory acts or behavior), 2 (aborted attempt), 3 (interrupted attempt), and 4 (actual attempt). More than 1 classification can be selected provided they represent separate episodes. (Minimum total score 0, maximum total score 5; higher total scores indicate more suicidal ideation and/or suicidal behavior)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (116):
- United States (42):
  - Duplicate_Barrow Neurological Institute /ID# 228217, Phoenix, Arizona
  - California Headache and Balance Center /ID# 226241, Fresno, California
  - Duplicate_Pharmacology Research Institute (PRI) - Los Alamitos (Wake) /ID# 226404, Los Alamitos, California
  - Pharmacology Research Institute (PRI) - Newport Beach (Wake) /ID# 226389, Newport Beach, California
  - Excell Research, Inc /ID# 228390, Oceanside, California
  - Duplicate_Schuster Medical Research Institute /ID# 226246, Sherman Oaks, California
  - Alpine Clinical Research Center /ID# 226203, Boulder, Colorado
  - Sensible Healthcare /ID# 226426, Ocoee, Florida
  - Accel Research Sites - Tampa Clinical Research Unit /ID# 226252, Tampa, Florida
  - NeuroTrials Research Inc /ID# 226477, Atlanta, Georgia
  - Allied Physicians - Fort Wayne Neurological Center /ID# 226390, Fort Wayne, Indiana
  - Josephson-Wallack-Munshower Neurology - Northeast /ID# 226295, Indianapolis, Indiana
  - Collective Medical Research /ID# 226482, Overland Park, Kansas
  - Ochsner Clinic Foundation /ID# 228220, Covington, Louisiana
  - Pharmasite Research, Inc. /ID# 226444, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center /ID# 228214, Boston, Massachusetts
  - BTC of New Bedford /ID# 226289, New Bedford, Massachusetts
  - Clinical Research Institute, Inc /ID# 226232, Minneapolis, Minnesota
  - Headache Neurology Research Institute /ID# 226234, Ridgeland, Mississippi
  - StudyMetrix Research /ID# 226296, City of Saint Peters, Missouri
  - Clinvest Research LLC /ID# 226275, Springfield, Missouri
  - Methodist Physicians Clinic/CCT Research /ID# 226422, Fremont, Nebraska
  - Albuquerque Clinical Trials, Inc. /ID# 226523, Albuquerque, New Mexico
  - Albany Medical Center Rheumatology /ID# 228212, Albany, New York
  - Headache Wellness Center /ID# 226233, Greensboro, North Carolina
  - Duplicate_CTI Clinical Research Center /ID# 226278, Cincinnati, Ohio
  - Stetson-University of Cincinnati /ID# 226326, Cincinnati, Ohio
  - Abington Neurological Associates - Abington /ID# 226449, Abington, Pennsylvania
  - Preferred Primary Care Physicians, Inc. /ID# 226447, Pittsburgh, Pennsylvania
  - Mount Vernon Clinical Research /ID# 226249, Chattanooga, Tennessee
  - CNS Healthcare - Memphis /ID# 226254, Memphis, Tennessee
  - FutureSearch Trials of Neurology /ID# 226424, Austin, Texas
  - Austin Clinical Trial Partners /ID# 228391, Austin, Texas
  - DiscoveResearch, Inc /ID# 226490, Bryan, Texas
  - Texas Neurology /ID# 226425, Dallas, Texas
  - LinQ Research, LLC /ID# 226391, Pearland, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic /ID# 226248, Salt Lake City, Utah
  - J. Lewis Research, Inc. Foothill Family Clinic South /ID# 226328, Salt Lake City, Utah
  - Highland Clinical Research /ID# 226287, Salt Lake City, Utah
  - Sentara Family Medicine Physicians /ID# 226448, Virginia Beach, Virginia
  - Northwest Clinical Research Center /ID# 226240, Bellevue, Washington
  - Puget Sound Neurology /ID# 226253, Tacoma, Washington
- Canada (5):
  - CHAMP Clinic /ID# 226256, Calgary, Alberta
  - Vancouver Island Health Authority /ID# 226255, Victoria, British Columbia
  - Aggarwal and Associates Limited /ID# 226452, Brampton, Ontario
  - Ottawa Headache Centre Research Inc /ID# 226451, Ottawa, Ontario
  - Diex Recherche Sherbrooke Inc. /ID# 226427, Sherbrooke, Quebec
- Czechia (13):
  - CCR Ostrava, s.r.o. /ID# 228412, Ostrava, Ostrava-mesto
  - A-Shine s.r.o. /ID# 226207, Pilsen, Plzeň Region
  - NeuroHK s.r.o. /ID# 226429, Hradec Králové
  - BRAIN-SOULTHERAPY s.r.o. /ID# 226394, Kladno
  - Pratia Pardubice a.s. /ID# 226393, Pardubice
  - Clintrial s.r.o. /ID# 228413, Prague
  - DADO MEDICAL s.r.o. /ID# 226421, Prague
  - Pratia Prague s.r.o. /ID# 226406, Prague
  - Fakultni Thomayerova nemocnice /ID# 228409, Prague
  - FORBELI s.r.o. /ID# 228406, Prague
  - INEP medical s.r.o. /ID# 228411, Prague
  - Vestra Clinics s.r.o. /ID# 226453, Rychnov nad Kněžnou
  - NeuroMed Zlin s.r.o. /ID# 228414, Zlín
- Rigshospitalet Glostrup /ID# 228417, Glostrup Municipality, Capital Region, Denmark
- France (6):
  - CHU Nice - Hopital de Cimiez /ID# 228419, Nice, Alpes-Maritimes
  - AP-HM - Hopital de la Timone /ID# 226407, Marseille, Bouches-du-Rhone
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord /ID# 228418, St-Priest-en-Jarez, Pays de la Loire Region
  - Duplicate_Hôpital Pierre Wertheimer /ID# 226430, Bron, Rhone
  - CHU Clermont Ferrand - Hopital Gabriel Montpied /ID# 226459, Clermont-Ferrand
  - AP-HP - Groupe Hospitalier 10e - Hopital Lariboisiere /ID# 226220, Paris
- Germany (11):
  - Neuropoint GmbH /ID# 226313, Ulm, Baden-Wurttemberg
  - Neuropraxis Muenchen Sued /ID# 226309, Unterhaching, Bavaria
  - Klinische Forschung Hannover-Mitte GmbH /ID# 226305, Hanover, Lower Saxony
  - Studienzentrum Nord-West /ID# 226310, Westerstede, Lower Saxony
  - AmBeNet GmbH /ID# 226312, Leipzig, Saxony
  - Schmerzklinik Kiel /ID# 226454, Kiel, Schleswig-Holstein
  - Zentrum für Neurologie, Neurochirurgie und Psychiatrie /ID# 229991, Berlin
  - Praxis Dr. Gendolla /ID# 229988, Essen
  - Universitaetsklinikum Essen /ID# 229989, Essen
  - Vitos Orthopaedische Klinik Kassel gemeinnuetzige GmbH /ID# 231571, Kassel
  - Velocity Clinical Research /ID# 226307, Wiesbaden
- Hungary (4):
  - Gyongyosi Bugat Pal Korhaz /ID# 228429, Gyöngyös, Heves County
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 226409, Kaposvár, Somogy County
  - Clinexpert Kft /ID# 228431, Budapest
  - S-Medicon Kft /ID# 228432, Budapest
- Italy (6):
  - Azienda Ospedaliero Universitaria Careggi /ID# 228624, Florence, Firenze
  - Ospedale Ss. Filippo e Nicola /ID# 228627, Avezzano, L Aquila
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 228625, Milan, Milano
  - IRCCS San Raffaele /ID# 228436, Rome, Roma
  - Universita di Pavia /ID# 228628, Pavia
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 228630, Roma
- Netherlands (2):
  - Canisius-Wilhelmina Ziekenhuis /ID# 226410, Nijmegen, Gelderland
  - ZorgSaam Zorggroep Zeeuws-Vlaanderen /ID# 226456, Terneuzen, Zeeland
- Poland (9):
  - Solumed Centrum Medyczne /ID# 226298, Poznan, Greater Poland Voivodeship
  - Vitamed Galaj i Cichomski Sp.j. /ID# 226416, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o. /ID# 228631, Krakow, Lesser Poland Voivodeship
  - Centrum Leczenia Padaczki i Migreny /ID# 226458, Krakow, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej /ID# 226412, Lublin, Lublin Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 226431, Gdynia, Pomeranian Voivodeship
  - Silmedic Sp. z o.o. /ID# 226457, Katowice, Silesian Voivodeship
  - EuroMedis sp. z o.o. /ID# 226413, Szczecin, West Pomeranian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak /ID# 226417, Wroclaw
- South Korea (7):
  - Duplicate_Pusan National University Hospital /ID# 231416, Busan, Busan Gwang Yeogsi
  - Hallym University Dongtan Sacred Heart Hospital /ID# 226264, Hwaseong, Gyeonggido
  - Nowon Eulji Medical Center, Eulji University /ID# 226261, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 226199, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 226263, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 226280, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 226265, Seoul
- Spain (4):
  - Duplicate_CLINICA UNIVERSIDAD DE NAVARRA-Pamplona /ID# 226335, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron /ID# 226338, Barcelona
  - Hospital Universitario Virgen del Rocio /ID# 226333, Seville
  - Hospital Clinico Universitario de Valladolid /ID# 226330, Valladolid
- Taiwan (4):
  - Kuang-Tien General Hospital /ID# 226259, Taichung, Taichung
  - Tainan Sin Lau Hospital /ID# 226229, Tainan, Tainan
  - Taipei Veterans General Hospital /ID# 226206, Taipei City, Taipei
  - Tri-Service General Hospital /ID# 228998, Taipei
- United Kingdom (2):
  - King's College Hospital NHS Foundation Trust /ID# 226524, London
  - Re:Cognition Health - London /ID# 231205, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Ashina S, Ashina M, Holle-Lee D, Tassorelli C, Cho SJ, He MY, De Abreu Ferreira R, Gandhi P, Smith JH, Pfleeger K, Trugman JM. Long-term safety, efficacy and functional outcomes of atogepant for the preventive treatment of migraine. Cephalalgia. 2025 Aug;45(8):3331024251365206. doi: 10.1177/03331024251365206. Epub 2025 Aug 19. PMID 40831083
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=3101-312-002